CLINICAL TRIAL: NCT04849832
Title: Evaluating the Effect of Polyphenols on the Iron Bioavailability From Iron Chlorophyllin in Young Women Using the Iron Stable Isotopic Method
Brief Title: Effect of Polyphenols on Absorption of Iron From Sodium Iron Chlorophyllin
Acronym: polySIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PolySIC
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Tea

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, single centre cross over study where every participant will receive all the four interventions.
Masking Description: There will be no masking as the ferrous sulfate solutions will be colourless compared to the green color solution of SIC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SIC (Experimental): 4mg of Fe will be given as 102 mg of SIC as a solution
  Interventions: Dietary Supplement: SIC
- SIC + tea (Experimental): 4 mg of Fe will be given as 102 mg of SIC as a solution along with 200 ml of black tea
  Interventions: Dietary Supplement: SIC + tea
- FeSO4 (Active Comparator): 4 mg of Fe will be given as Ferrous sulfate solution
  Interventions: Dietary Supplement: FeSO4
- FeSO4 + tea (Active Comparator): 4 mg of Fe will be given as Ferrous sulfate solution along with 200 ml of black tea
  Interventions: Dietary Supplement: FeSO4 + tea

INTERVENTIONS:
Dietary Supplement: SIC — Sodium Iron Chlorophyllin as prepared by the human nutrition laboratory, ETH Zurich
  Arms: SIC
Dietary Supplement: SIC + tea — Sodium Iron Chlorophyllin as prepared by the human nutrition laboratory, ETH Zurich with 2g of tea brewed for 5 minutes
  Arms: SIC + tea
Dietary Supplement: FeSO4 — Ferrous sulfate solution serves as a positive control - and whose absorption is well known.
  Arms: FeSO4
Dietary Supplement: FeSO4 + tea — Ferrous sulfate solution given with 2g of tea brewed for 5 minutes - expected iron absorption inhibition
  Arms: FeSO4 + tea

SUMMARY:
Polyphenols present in tea are known to inhibit the absorption of non heme iron. The inhibiting effect of tea on non-heme iron absorption is attributed to the flavonoids present in tea. It is well known that Ferrous sulfate is not absorbed well in the presence of polyphenols. We would like to evaluate the effect of polyphenols on the newly developed compound, sodium iron chlorophyllin (SIC), which mimics the heme iron structure. Comparisons of fractional absorption of SIC and Ferrous Sulfate in the presence of polyphenols can help identify the performance of the compounds as vehicles for iron delivery in the presence of iron absorption inhibitors.

In a single-blind randomized cross-over study using stable iron isotope technique, iron bioavailability from SIC delivered with an inhibitory matrix can therefore be determined when given along with black tea

DETAILED DESCRIPTION:
New approaches to treat iron deficiency include developing novel iron compounds with possible iron absorption routes that increase iron bioavailability and reduce gastrointestinal side effects.

Sodium iron chlorophyllin (SIC) is a water-soluble semisynthetic chlorophyll derivative where the magnesium in the porphyrin ring has been substituted by iron. Given the porphyrin ring heme-like structure of SIC, it may be an alternative delivery route for iron, suitable also for vegetarians and vegans. Yet, there are few studies investigating the use of SIC for this purpose.

We recently completed the study entitled "Evaluation of iron bioavailability from iron chlorophyllin in young women using the iron stable isotopic method" based on previous in vitro and in vivo studies.. The study showed a 7% fractional iron absorption (FIA) from SIC when compared to the control compound, ferrous sulfate, which had a FIA of 30%, indicating a Relative Bioavailability of SIC of 20%. The study showed an inverse relationship between ferritin status and iron absorption from SIC in the study participants and an increase in the FIA in the presence of ascorbic acid. Both these findings lean towards the possibility that that the iron contributing to the FIA from SIC may be iron that was dissociated from the porphyrin ring of the chlorophyllin and entering the common non heme iron pool. This inverse relationship in ferritin and FIA is well known for ferrous sulfate. However, one cannot confirm the pathway taken up by SIC to deliver iron based on the previous study alone.

Polyphenols present in tea are known to inhibit the absorption of non heme iron.The inhibiting effect of tea on non-heme iron absorption is attributed to the flavonoids present in tea. There are several types of tea flavonoids: monomers (catechin), dimers (theaflavin), and polymers (thearubigin). Black tea contains 10% flavanols, 25% catechins, 20% theaflavins and 45% thearubigins. The mechanism of iron absorption inhibition by tea is by formation of a complex of the flavonoids with iron. It is mainly the galloyl group in these phenolic compounds that specifically binds iron. A cup of black tea, brewed with 2.5 g tea leaves contains about 200 mg tea flavonoids . Heme iron absorption has also been shown to be inhibited by the presence of polyphenols but unclear to what extent. Thus, comparisons of fractional absorption of SIC and Ferrous Sulfate in the presence of polyphenols can help identify the performance of the compounds as vehicles for iron delivery in the presence of iron absorption inhibitors.

In a single-blind randomized cross-over study using stable iron isotope technique, iron bioavailability from SIC delivered with an inhibitory matrix can therefore be determined when given along with black tea.

SIC has been produced at the HNL with a 50% incorporation of iron into the chlorophyll. Our protocol is based on a Unilever patent that is no longer active, with in-house adaptation. The SIC has a neutral taste and will be presented as a dark green liquid, being the solution of SIC in water.

If SIC, as hypothesized, behaves in a similar way to heme, then iron absorption inhibitors, such as the polyphenols, will not have an effect on the absorption of iron from SIC.

ELIGIBILITY:
Inclusion Criteria:

* female aged between 18-45 y old;
* SF <80 µg/L;
* BMI 18.5-24.9 kg/m2;
* weight <70 kg;
* signed informed consent;
* able to communicate and comprehend English language.

Exclusion Criteria:

* anemia (Hb <12 g/dL);
* Inflammation (CRP > 5 mg/L);
* chronic digestive, renal and/or metabolic disease;
* chronic medications (except for oral contraceptives);
* use of vitamin, mineral and pre- and/or probiotic supplements in the previous 2 weeks before study initiation and during the course of the study;
* blood transfusion, blood donation or significant blood loss over the past 4 months;
* difficulties with blood sampling;
* antibiotic treatment in the 4 weeks before study initiation;
* pregnancy (tested in serum at screening) or intention to become pregnant;
* lactation up to 6 weeks before study initiation;
* earlier participation in a study using stable isotopes or participation in any clinical study within the last 30 days;
* unable to comply with study protocol (e.g. not available on certain study appointment days or difficulties with blood withdrawal);
* inability to understand the information sheet and the informed consent form due to cognitive or language reasons;
* smoking;
* unwilling to use an effective method of contraception.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females
Enrollment: 40 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Ratio of FIA of SIC arms vs ratio of FIA of Ferrous sulfate arms | Day 1 of the study
  ratio of iron bioavailability (as measured by erythrocyte incorporation of the stable isotope labels) from SIC in a polyphenol matrix to that from SIC alone with the ratio of iron bioavailability from FeSO4 in a polyphenol matrix to that from FeSO4 alone.
Ratio of FIA of SIC arms vs ratio of FIA of Ferrous sulfate arms | Day 17 of the study
  ratio of iron bioavailability (as measured by erythrocyte incorporation of the stable isotope labels) from SIC in a polyphenol matrix to that from SIC alone with the ratio of iron bioavailability from FeSO4 in a polyphenol matrix to that from FeSO4 alone.
Ratio of FIA of SIC arms vs ratio of FIA of Ferrous sulfate arms | Day 33 of the study
  ratio of iron bioavailability (as measured by erythrocyte incorporation of the stable isotope labels) from SIC in a polyphenol matrix to that from SIC alone with the ratio of iron bioavailability from FeSO4 in a polyphenol matrix to that from FeSO4 alone.

SECONDARY OUTCOMES:
Hemoglobin | day 1, day 17 and day 33 of the the study
  Iron status biomarker
Ferritin | day 1, day 17 and day 33 of the the study
  Iron status biomarker
sTfR | day 1, day 17 and day 33 of the the study
  Iron status biomarker
C-reactive Protein | day 1, day 17 and day 33 of the the study
  Inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Farebrother, Dr.Sc, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zürich, Laboratory of Human Nutrition, Zurich, Canton of Zurich, Switzerland